CLINICAL TRIAL: NCT04956926
Title: An Open-label, First-in-human, Dose Escalation and Expansion Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of JS201 in Patients With Advanced Malignant Tumors
Brief Title: Clinical Study of JS201 in Patients With Advanced Malignant Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS201-001-I
Record Dates: First submitted 2021-06-23; First posted 2021-07-09 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2021-08

CONDITIONS: Patients With Advanced Malignant Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS201 (Experimental)
  Interventions: Drug: JS201

INTERVENTIONS:
Drug: JS201 — JS201 is administered intravenously Q3W at the corresponding dose.

SUMMARY:
This is an open label, phase I clinical study to evaluate the safety, tolerability, pharmacokinetic (PK) profile, pharmacodynamic (PD) profile, immunogenicity and preliminary efficacy of JS201 in the patients with advanced malignant tumors who have progression after or during the standard of care, or no effective standard therapeutic regimen. This study is divided into three phases: dose-escalation phase, dose expansion phase, and clinical expansion phase.

ELIGIBILITY:
Inclusion Criteria

1. Understanding and voluntarily signing the informed consent form;
2. Male or female, aged 18 to 70 years (inclusive), for the dose-expansion and clinical expansion parts, aged 18 to 75 years (inclusive);
3. Patients with histologically or cytologically confirmed advanced malignant tumors who have progression after or on the standard of care, or have no effective standard therapeutic regimen;
4. In the clinical expansion stage, patients with advanced cervical cancer, lymphoma, non-small cell lung cancer (NSCLC), gastric cancer, urothelial cancer and other malignant solid tumors diagnosed by histology or cytology were enrolled (the details shown in the full protocol);
5. ECOG PS score: 0~1;
6. Patients with life expectancy ≥12 weeks;
7. At least one measurable lesion per RECIST v1.1 (solid tumors) or 2014 Lugano (lymphoma) criteria;
8. Agree to provide fresh biopsies prior to first dose, or archived samples within two years if there is unpredictable risk of biopsy to the patient（at least 15 fresh biopsy sections or 11 surgical sections). For patients who cannot provide abovementioned sections of tissue samples due to special conditions, it needs to contact with the medical monitor of the sponsor to confirm whether this inclusion criterion can be exempted;
9. Function of vital organs must meet the followings (no blood transfusion or hematopoietic stimulating factor used within 14 days prior to the first dose

   Absolute neutrophil count (ANC) ≥1.5×109/L;

   Platelet (PL) ≥100×109/L;

   Hemoglobin (Hb) ≥ 9 g/dL;

   Total bilirubin (TBIL) ≤1.5 × ULN; if there is hepatic metastasis, total bilirubin ≤2 × ULN; direct bilirubin (dBIL) ≤ 3.0mg/dL in the patients with Gilbert's syndrome;

   Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN; or ≤5 × ULN in the patients with hepatic metastasis;

   Serum creatinine (Cr) ≤1.5 × ULN, or calculated creatinine clearance (using Cockcroft -Gault formula) ≥50 mL/min, or 24-hour urine creatinine clearance ≥ 50 mL/min;

   International normalized ratio (INR) ≤1.5 × ULN and activated partial thromboplastin time (aPTT) ≤1.5 × ULN in the patients receiving no anticoagulation therapy;

   QTc interval ≤450 ms for man and ≤470 ms for woman, as calculated using Fridericia's formula;
10. Female patients of childbearing potential and male patients with partners of childbearing potential must agree to use a medically recognized contraceptive measure (e.g., intrauterine device IUD, contraceptive or condom) during the study and within 3 months after the end of treatment; the serum HCG test must be negative in the female patients with childbearing potential within 7 days prior to enrollment; and the female patients must be not lactating.

Exclusion criteria

1. Known allergy to any component of JS201;
2. The patients have previously received the TGF-β/TGF-β receptor targeted drugs;
3. Received other investigational product within 4 weeks prior to the first dose of JS201;
4. Accepted major surgery (judged by investigator) or in the recovery period of the surgery within 4 weeks after the first dose of JS201;
5. Antitumor chemotherapy (6 weeks after the last dose of nitrosourea or mitomycin chemotherapy), radiotherapy, hormone therapy, targeted therapy (for small molecular targeted therapy, within 2 weeks prior to the first dose of JS201), immunotherapy (e.g., anti-PD1/PD-L1 and anti-CTLA-4 therapy) or biotherapy (e.g., cell therapy) within 4 weeks prior to the first dose. Local palliative therapy for isolated lesion is acceptable (e.g., local surgery or radiotherapy), if the tumor evaluation is not affected;
6. Use of immunosuppressive drug or immune enhancing drugs (such as thymosin, interferon, interleukin, etc.) within 2 weeks prior to the first dose. However, corticosteroid nasal spray, inhaler or ≤10 mg/day systemic prednisone and equivalent similar products are accepted. Short-term use of systemic corticosteroid therapy with a dose equivalent to prednisone > 10 mg / day (e.g. for the treatment/prevention of contrast medium allergy) with ≤ 3 days is allowed;
7. Previous allogeneic bone marrow transplantation or solid organ transplantation;
8. Live attenuated vaccine within 30 days prior to the first dose is excluded, and inactivated influenza vaccination is allowed;
9. Having other malignant tumor other than the disease investigated within 5 years prior to the first dose. The malignant tumors, including but not limited to sufficiently treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell carcinoma of skin, or ductal carcinoma in situ treated with radical surgery, are eligible;
10. Symptomatic central nervous system (CNS) metastasis requiring intervention (including corticosteroids and antiepileptics). Asymptomatic CNS metastasis previously treated with local therapy is eligible. If the patients confirmed CNS metastasis during screening without any symptoms, and no intervention is required per the standard of care, the eligibility should be determined with the medical monitor of the sponsor;
11. No remission from the toxicity of previous antitumor therapy, i.e., not resolved to baseline, grade 0-1 per NCI-CTCAE v5.0 (except alopecia) or the level specified in the inclusion/exclusion criteria. Patients with irreversible toxicity reasonably expected to be non-aggravated by the study drug (e.g., hearing loss) can participate in this study upon discussion with the medical monitor of the sponsor;
12. Patients have accepted anti PD-1/PD-L1 monoclonal antibody treatment, and immune related adverse events occurred that stop the treatment;
13. Massive pleural effusion, ascites or pericardial effusion with clinical symptoms or requiring symptomatic treatment;
14. Active autoimmune disease requiring systemic therapy (e.g., corticosteroids or immunosuppressants) within 2 years prior to the first dose.

1) The autoimmune diseases include but not limited to systemic lupus erythematosus, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism and multiple sclerosis;

2) Patients with leukoderma or childhood asthma that has been completely relieved and does not need any intervention in adulthood can be enrolled;

3) For the patients combined with rheumatoid arthritis and other joint diseases, Sjogren's syndrome, celiac disease and psoriasis that have been controlled after local therapy, as well as those with positive antinuclear antibody (ANA) and antithyroid antibody, it should be evaluated whether the target organ is involved and systemic treatment is needed, and their enrollment will be determined by investigator;

4) Replacement therapy (e.g., thyroxine, insulin or physiological dose of corticosteroid for adrenal or pituitary insufficiency) will not be regarded as systemic treatment;

5) Patients requiring intermittent use of bronchodilators, inhaled corticosteroids or local injection of corticosteroids for chronic obstructive pulmonary disease (COPD) and asthma can be enrolled.

15. Active infection requiring systematic treatment/antibiotics or intravenous use of systemic anti-infection therapy with 1 week prior to the first dose or use for more than 7 days;

16. History of concurrent serious cerebro- and cardiovascular diseases: ≥grade 3 symptomatic congestive heart failure in accordance with New York Heart Association (NYHA) cardiac function grading system, poorly controlled hypertension or arrhythmia, unstable angina pectoris, myocardial infarction, cerebrovascular accident or transient ischemic attack within 6 months prior to the first doses, or any other arterial thrombosis or embolic event;

17. Presence of active tuberculosis, or interstitial lung disease requiring oral or intravenous steroids or history of pneumonia;

18.Hepatitis (nonalcoholic steatohepatitis and alcoholic/drug-related/autoimmune hepatitis) or cirrhosis;

19. Known positive for human immunodeficiency virus (HIV);

20. Patients with evidence of active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients with HBcAb positive and/or HBsAg positive in the screening stage, if the patients with HBV DNA copy number < 1000 CPS/ml or < 200 IU/ml can be enrolled. HBsAg positive patients must receive antiviral treatment throughout the study period. Patients with positive HCV antibody in the screening stage can be recruited only when the HCV RNA test result is negative;

21. Any other clinical significant diseases or conditions can effect on the compliance with the protocol (e.g., history of psychosis or drug abuse), the signature of the informed consent form (e.g., drug addiction and drug abuse), or is unsuitable to be involved in this clinical trial, which determined by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2021-07-29 (Actual); Primary Completion 2023-07-07 (Estimated); Study Completion 2023-07-07 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with DLT (Dose limiting Toxicity) | 21 days after first infusion of study drug
  DLT is defined as any of the specified toxicities evaluated as at least possibly related with the study drug within 21 days after the first dose (NCI-CTCAE v5.0);
Number of Subjects with adverse event (AE) | Up to 2 years
  An Adverse Event (AE) is defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship.
Number of Subjects with serious adverse event (SAE) | Up to 2 years
  A Serious Adverse Event (SAE) is an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect
Number of Subjects with immune related adverse event (irAE) | Up to 2 years
  IrAE is assessed according to the judgement of investigators

SECONDARY OUTCOMES:
anti-drug body (ADA) | Up to 2 years
  incidence of anti-drug body (ADA)
peak concentration (Cmax) | Up to 2 years
  Cmax after JS201 administration
trough concentration (Ctrough) | Up to 2 years
  Ctrough after JS201 administration
area under the plasma drug concentration-time curve (AUC0-t ) | Up to 2 years
  AUC0-t after JS201 administration
volume of distribution (Vss) | Up to 2 years
  Vss after JS201 administration
elimination half-life (t1/2) | Up to 2 years
  t1/2 after JS201 administration
clearance rate (CL) | Up to 2 years
  CL after JS201 administration
ORR | Up to 2 years
  The efficacy evaluated by the investigator in accordance with RECIST 1.1 criteria (solid tumors) or Lugano criteria (2014, lymphoma), including complete response (CR) and partial response (PR).
DOR | Up to 2 years
  DOR is defined as the time from the date of the first documentation of response (confirmed CR or confirmed PR) to the date of the first documentation of PD or death due to any cause, whichever occurs first.
DCR | Up to 2 years
  The efficacy evaluated by the investigator per RECIST 1.1 criteria (solid tumors) or Lugano criteria (2014, lymphoma), including CR, PR and stable disease (SD);
PFS | Up to 2 years
  PFS is defined as the time from the date of randomization to the earlier of the dates of the first documentation of progressive disease or death due to any cause.
OS | Up to 2 years
  OS is defined as the time from the date of randomization to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Beiijng Cancer Hospital, Beijin, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangong
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Harbin medical University cancer hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhenzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Techonoly, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shandong Tumor Hospital, Jinan, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Cancer Hospital of the University of Chinese Academy of Sciences, Hangzhou, Zhejiang
  - Sun Yat-sen University Cancer Center, Guangzhou